CLINICAL TRIAL: NCT03337958
Title: Evaluation of an Educational Intervention in the Management of Inhalers With Tablet and Ventilatory Reeducation: a Randomized Clinical Study
Brief Title: Education With Inhalers in Patients With COPD Exacerbation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Principal investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DF0071UG
Record Dates: First submitted 2017-09-20; First posted 2017-11-09 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Education; Dry Powder Inhalers; Metered Dose Inhalers; Pulmonary Disease; Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL GROUP (No Intervention): Received the standard medical and pharmacological care provided by the hospital
- INTERVENTION GROUP (Experimental): The group received the standard medical and pharmacological care provided by the hospital. In addition, an educational program on the use of inhalers, which included an explanation of the use of inhalers together with a ventilatory re-education program, furthermore, the technique of inhaler use was trained.
  Interventions: Device: Ventilatory re-education

INTERVENTIONS:
Device: Ventilatory re-education — The first day of intervention consisted primarily in ventilatory re-education. During the realization of the technique he was videotaped with a Tablet so that later the patient could be seen and on the video to be able to give him the guidelines for the correction. On the second and third day of the intervention, ventilation re-education was performed and the inhalation technique was subsequently trained.
  Arms: INTERVENTION GROUP

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a public health problem with great morbidity. The main therapeutic strategy is inhalers. The objective of this study is to determine the efficacy of an educational intervention in the use of inhalers in patients with COPD including ventilatory re-education and video recordings of the patients themselves.

DETAILED DESCRIPTION:
The importance of this pathology lies not only in its high prevalence, which is expected to increase due to the aging of society but also in its high mortality. In Europe, it is estimated that 50% of adult patients do not use the inhaler correctly. The clinical development of COPD includes periods of stability interspersed with symptomatic exacerbations, which usually involve hospitalization. During these hospitalizations, respiratory symptoms are worsening.Nevertheless, in Europe, it is estimated that 50% of adult patients do not use the inhaler correctly. Thus, it is very important the pharmacological education in this patients.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were to be clinically diagnosed of exacerbation of COPD, to possess pharmacological treatment in the form of inhalers.

Exclusion Criteria:

* Exclusion criteria were inability to provide informed consent, presence of psychiatric or cognitive disorders, neurological disorders, organ failure, cancer or inability to cooperate. Patients who had experienced an exacerbation of prior COPD in less than one month were excluded.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Respiratory parameters | baseline, 12 months
  Changes from baseline to postintervention in respiratory parameters using a spirometer. The most important respiratory parameters evaluated is forced expiratory volume in the first second (FEV1)

SECONDARY OUTCOMES:
Knowledge of the disease | Baseline, 12 months
  Evaluated at baseline by EPOC-Q
Cognitive Level | Baseline
  Cognitive level was assessed using the Montreal Cognitive Assessment (MOCA).
Functional independence | Baseline
  Functional independence was assessed using the Functional Independence Scale (FIM).
Anxiety-depression level | Baseline
  Changes from baseline to postintervention in anxiety and depression measured with the Hospital Anxiety and Depression Scale. Patients are going to complete this questionnaire composed of statements relevant to either generalized anxiety or depression.
Adhesion to inhalers | Baseline
  Level of adhesion to inhalers was assessed with TAI (Inhaler Adhesion Test).
Dyspnea level | baseline, 12 months
  Perceived perception of dyspnea was collected through the Modified Borg Scale.
Physical fitness | baseline, 12 months
  Physical fitness was assessed by performing the five-times-sit-to-stand test. It consists of getting up and sitting five times in a row without a support. The time period in which the exercise is performed is the patient's score with a maximum of 60 seconds.
Technique of the inhaler | baseline, 12 months
  The evaluation of the technique of the inhalers was carried out by means of a checklist composed of 5 items. Checked those points that were done correctly obtaining 5 points if the technique that was done correctly.
Respiratory parameters | baseline, 12 months
  Changes from baseline to postintervention in respiratory parameters using a spirometer as recommended by the American Thoracic Society. The most important respiratory parameters evaluated are forced vital capacity (FVC), carbon dioxide partial pressure (PCO2) and oxygen partial pressure (PO2).

CONTACTS AND LOCATIONS:
Overall Officials: Marie Carmen Valenza, PT, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Department of Physical Therapy, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided